CLINICAL TRIAL: NCT05109130
Title: Sixth Affiliated Hospital, Sun Yat-sen University
Brief Title: Change of Circulating Tumor Cells During Laparoscopic or Transanal Endoscopic Surgery for Rectal Cancer.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Sun Yat-sen University, Sun Yat-sen University
Other Study IDs: GIHSYSU-20
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Rectal Neoplasms; Neoplastic Cells, Circulating; Laparoscopic Surgery; Transanal Endoscopic Surgery
Keywords: rectal cancer; CTCs
MeSH Terms: conditions — Rectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic surgery: Laparoscopic total mesorectal excision was performed on the enrolled patients.
  Interventions: Procedure: Surgical approach
- Transanal endoscopic surgery: Transanal total mesorectal excision was performed on the enrolled patients.
  Interventions: Procedure: Surgical approach

INTERVENTIONS:
Procedure: Surgical approach — Different surgical methods for rectal cancer resection

SUMMARY:
The primary purpose of this study is to compare the changes of circulating tumor cells (CTCs) at different time points in rectal cancer patients undergoing laparoscopic or transanal endoscopic radical resection. Our secondary purpose is to explore the effects of perioperative circulating tumor cells on tumor recurrence and metastasis.

DETAILED DESCRIPTION:
Mid-low rectal cancer is one of the common malignant tumors and the incidence has increased significantly in recent years. At present, surgery is still the most important and effective method for the treatment of mid-low rectal cancer. Traditional laparoscopic surgery and emerging transanal total mesorectal excision (TaTME) are the main methods. More than one-third of rectal cancer patients will eventually occur local recurrence and distant metastasis, which are the most important factors affecting prognosis. Circulating tumor cells may lead to distant metastasis, so the detection of CTCs in blood has important clinical significance in predicting the recurrence and metastasis of rectal cancer and monitoring treatment response. Due to the different degrees of contact between distinct surgical methods, this may lead to an increase in the quantity of CTCs in the blood, which may affect the prognosis of patients. Therefore, the investigators conducted a randomized controlled study to compare the changes in the quantity of CTCs in the central vein before, during and after operation in rectal cancer patients undergoing transanal endoscopic or laparoscopic radical resection. To explore the effect of two surgical methods on the risk of micrometastasis, and to provide evidence for the selection and improvement of rectal cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Mid-low rectal cancer.
2. Single lesion.
3. No metastasis.
4. Clinical Stage T2-3, N0-1.

Exclusion Criteria:

1. History of malignant tumors.
2. Acute bowel obstruction, bleeding or perforation.
3. Received neoadjuvant treatment.
4. Tumor over 6cm in diameter or in severe adhesion with surrounded tissues.
5. Severe other contradictions of surgery.
6. Pregnant women will be excluded.

Exit Criteria:

1. The patient suffered from massive hemorrhage.
2. The operation mode needs to be changed according to the patient's condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 rectal cancer patients will be enrolled. Patients must be older than 18 years.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Change of circulating tumor cells during laparoscopic or transanal endoscopic surgery | 1 years
  To determine the changes of circulating tumor cells in rectal cancer patients undergoing laparoscopic or transanal endoscopic radical resection before operation and 5 days after operation.

SECONDARY OUTCOMES:
Disease free survival | 3 years
  Determine relationship of CTC numbers and local recurrence and distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Liang Huang, Principal Investigator — Sun Yat-sen University Sixth Affiliated Hospital
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided